CLINICAL TRIAL: NCT00669721
Title: Effects of UFH and LMWH on Osteoprotegerin and RANKL Plasma Levels in Hemodialysis Patients
Brief Title: OPG and RANKL Plasma Level After Administration of Unfractionated Heparin (UFH) and Low-Molecular-Weight Heparin (LMWH) in Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Prof. Sergio Stefoni, St. Orsola University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LWH-INT-79
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Renal Failure; Hemodialysis
Keywords: osteoprotegerin; RANKL; heparin; hemodialysis; anticoagulation; vascular calcification
MeSH Terms: conditions — Renal Insufficiency; Vascular Calcification | interventions — Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): This patients start a run in period with LMWH schedule as hemodialysis circuit anticoagulation. Then they'll undergo hemodialysis with LMWH for a second period of two weeks: in this checking phase samples will be collected during the midweek hemodialysis sessions. After the checking phase the patients will be crossed to UFH schedule. A wash out period of two weeks with UFH will be done. At the end of this period two weeks of checking phase will starts.
  Interventions: Drug: law molecular weigth heparin
- B (Active Comparator): The patients randomized to receive UFH will start a run in period with this heparin schedule. Then they'll undergo hemodialysis with UFH for a second period of two weeks: in this checking phase samples will be collected during the midweek hemodialysis sessions. After the checking phase the patients will be crossed to LMWH. A wash out period of two weeks with UFH will be done. At the end of this period two weeks of checking phase will starts.
  Interventions: Drug: unfractioned heparin

INTERVENTIONS:
Drug: law molecular weigth heparin — administration of LMWH as anticoagulation for hemodialysis circuit;nadroparin is administred ad the dosage of 65 IU/kg on starting dialysis and in the arterial hemodialytic line after a washing phase with 2 litres of a heparin-free saline solution 0.9%.
  Other Names: nadroparin
  Arms: A
Drug: unfractioned heparin — administration of UFH as anticoagulation of hemodialysis circuit; standard heparin ( Sodic Heparin, Vister by Parke-Davis) 1500 IU on starting dialysis and 1500 ± 500 IU in continues intradialytic infusion per dialysis session
  Other Names: standard heparin, Sodic Heparin
  Arms: B

SUMMARY:
A randomised, prospective, cross over study will be done to determine whether the anticoagulation therapy with UFH or LMWH used for hemodialysis sessions modifies osteoprotegerin and RANKL plasma levels.

DETAILED DESCRIPTION:
It's well known that treatment with heparin can lead to a reduction in bone density and the development of osteoporosis [ 1 ]. Until now, it's not clear the mechanism by which heparin produces this side effect, but several studies in animals [ 2,3] and in humans [ 4 ] have shown that LMWH may induce less osteoporosis than UFH.

Recently it was observed that heparin interferes with RANK/RANKL/POG system [5,6]. RANK, RANKL and OPG are members of TNF alfa receptor superfamily. The pathways involving them in conjunction with various cytokines and calciotrophic hormones play a pivotal role in bone remodelling. In addiction experimental and clinical studies established a consistent relationship between the RANK/RANKL/OPG pathway and both skeletal lesion related to disorders of mineral metabolism [7,8,9] and vascular calcification [7,10]. OPG exists either as active soluble form or is expressed by osteoblast, stromal and cardiovascular cells, acting as decoy receptor that competes with RANKL for RANK.

This interaction inhibits osteoclastic proliferation and differentiation and consequently prevents bone resorption . OPG is also produced by both endothelial cells (EC) and Vascular Smooth Muscle Cells (VSMCs ). EC-derived OPG seems to act as an important autocrine / paracrine factor able to protect against arterial calcification blocking the effects of RANKL that promotes monocytes differentiation in osteoclast -like cells and an osteogenic differentiation program in VSMC. This process leads to the synthesis of bone proteins and matrix calcification within the arterial vessel. OPG levels increase with aging and are higher in ESRD patient [11,12].

Recently it was demonstrated in cultures of murine bone marrow that the heparin inhibits osteoprotegerin activity binding OPG competitively and in this way inhibiting the interaction between OPG and RANKL [5].

On the other side heparin seems cause the mobilization of OPG into the circulation. It was reported that OPG is co-localized with vWF in Weibel Palade bodies in endothelial cells [13] and binds to Glucosaminoglycans (GAGs) at cellular membranes through its highly basic heparin binding domain [14,15]. Heparin treatment causes an immediate mobilization of these protein in to the circulation by displacement from the endothelial surface since they have higher affinity for heparins than GAGs at the endothelial surface[16,17]. UFH cause a more pronounced vascular mobilization of OPG than LMWH, indicating that UFH have an higher affinity for OPG than LMWH [6].

ELIGIBILITY:
Inclusion Criteria:

1. hemodialysis patients with age > 18 years on regular bicarbonate hemodialysis or hemodiafiltration treatment three times a week;
2. clinical stability at least three months before the study started;

Exclusion Criteria:

1. active gastrointestinal bleeding (one ore more positive hemoccult test in the last 8 weeks, melena or proctoraggia in the last 6 months )
2. hemorrhagic stroke
3. Myeloproliferative disorders
4. Hereditary deficiency of coagulation factors, LAC phenomenon or antiphospholipid syndrome
5. Malignant disease
6. Patient submitted to antithrombotic prophylaxis with LMWH
7. Immunosuppressive therapy
8. Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Levels of osteoprotegerin after administration of UFH or LMWH used as anticoagulant therapy for hemodialysis | during and after dialysis sessions

SECONDARY OUTCOMES:
Secondary aim of the study is to verify the safety of anticoagulation therapy with UFH and LMWH. | during and after dialysis sessions

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Stefoni, Prof, Principal Investigator — St.orsola University Hospital
Locations (1):
- St.Orsola University Hospital, Bologna, Italy

REFERENCES:
- [Background] Muir JM, Hirsh J, Weitz JI, Andrew M, Young E, Shaughnessy SG. A histomorphometric comparison of the effects of heparin and low-molecular-weight heparin on cancellous bone in rats. Blood. 1997 May 1;89(9):3236-42. PMID 9129028
- [Background] Pettila V, Leinonen P, Markkola A, Hiilesmaa V, Kaaja R. Postpartum bone mineral density in women treated for thromboprophylaxis with unfractionated heparin or LMW heparin. Thromb Haemost. 2002 Feb;87(2):182-6. PMID 11858475
- [Background] Irie A, Takami M, Kubo H, Sekino-Suzuki N, Kasahara K, Sanai Y. Heparin enhances osteoclastic bone resorption by inhibiting osteoprotegerin activity. Bone. 2007 Aug;41(2):165-74. doi: 10.1016/j.bone.2007.04.190. Epub 2007 May 5. PMID 17560185
- [Background] Vik A, Brodin E, Sveinbjornsson B, Hansen JB. Heparin induces mobilization of osteoprotegerin into the circulation. Thromb Haemost. 2007 Jul;98(1):148-54. PMID 17598007
- [Background] Collin-Osdoby P. Regulation of vascular calcification by osteoclast regulatory factors RANKL and osteoprotegerin. Circ Res. 2004 Nov 26;95(11):1046-57. doi: 10.1161/01.RES.0000149165.99974.12. PMID 15564564
- [Background] Vega D, Maalouf NM, Sakhaee K. CLINICAL Review #: the role of receptor activator of nuclear factor-kappaB (RANK)/RANK ligand/osteoprotegerin: clinical implications. J Clin Endocrinol Metab. 2007 Dec;92(12):4514-21. doi: 10.1210/jc.2007-0646. Epub 2007 Sep 25. PMID 17895323
- [Background] Orita Y, Yamamoto H, Kohno N, Sugihara M, Honda H, Kawamata S, Mito S, Soe NN, Yoshizumi M. Role of osteoprotegerin in arterial calcification: development of new animal model. Arterioscler Thromb Vasc Biol. 2007 Sep;27(9):2058-64. doi: 10.1161/ATVBAHA.107.147868. Epub 2007 Jul 5. PMID 17615383
- [Background] Nitta K, Akiba T, Uchida K, Otsubo S, Takei T, Yumura W, Kabaya T, Nihei H. Serum osteoprotegerin levels and the extent of vascular calcification in haemodialysis patients. Nephrol Dial Transplant. 2004 Jul;19(7):1886-9. doi: 10.1093/ndt/gfh263. Epub 2004 May 5. PMID 15128884
- [Background] Schoppet M, Shroff RC, Hofbauer LC, Shanahan CM. Exploring the biology of vascular calcification in chronic kidney disease: what's circulating? Kidney Int. 2008 Feb;73(4):384-90. doi: 10.1038/sj.ki.5002696. Epub 2007 Nov 28. PMID 18046319
- [Background] Zannettino AC, Holding CA, Diamond P, Atkins GJ, Kostakis P, Farrugia A, Gamble J, To LB, Findlay DM, Haynes DR. Osteoprotegerin (OPG) is localized to the Weibel-Palade bodies of human vascular endothelial cells and is physically associated with von Willebrand factor. J Cell Physiol. 2005 Aug;204(2):714-23. doi: 10.1002/jcp.20354. PMID 15799029
- [Background] Standal T, Seidel C, Hjertner O, Plesner T, Sanderson RD, Waage A, Borset M, Sundan A. Osteoprotegerin is bound, internalized, and degraded by multiple myeloma cells. Blood. 2002 Oct 15;100(8):3002-7. doi: 10.1182/blood-2002-04-1190. PMID 12351414
- [Background] Theoleyre S, Kwan Tat S, Vusio P, Blanchard F, Gallagher J, Ricard-Blum S, Fortun Y, Padrines M, Redini F, Heymann D. Characterization of osteoprotegerin binding to glycosaminoglycans by surface plasmon resonance: role in the interactions with receptor activator of nuclear factor kappaB ligand (RANKL) and RANK. Biochem Biophys Res Commun. 2006 Aug 25;347(2):460-7. doi: 10.1016/j.bbrc.2006.06.120. Epub 2006 Jun 30. PMID 16828054
- [Background] Valentin S, Larnkjer A, Ostergaard P, Nielsen JI, Nordfang O. Characterization of the binding between tissue factor pathway inhibitor and glycosaminoglycans. Thromb Res. 1994 Jul 15;75(2):173-83. doi: 10.1016/0049-3848(94)90066-3. PMID 7974391
- [Background] Hansen JB, Sandset PM, Huseby KR, Huseby NE, Nordoy A. Depletion of intravascular pools of tissue factor pathway inhibitor (TFPI) during repeated or continuous intravenous infusion of heparin in man. Thromb Haemost. 1996 Nov;76(5):703-9. PMID 8950777
- [Result] Deruelle P, Coulon C. The use of low-molecular-weight heparins in pregnancy--how safe are they? Curr Opin Obstet Gynecol. 2007 Dec;19(6):573-7. doi: 10.1097/GCO.0b013e3282f10e33. PMID 18007136
- [Result] Folwarczna J, Sliwinski L, Janiec W, Pikul M. Effects of standard heparin and low-molecular-weight heparins on the formation of murine osteoclasts in vitro. Pharmacol Rep. 2005 Sep-Oct;57(5):635-45. PMID 16227647
- [Result] Vescini F, Buffa A, Sinicropi G. Osteoprotegerina RANKL e RANK nella regolazione dell'ostoclastogenesi. Riv It Biol Med 22: 64-67, 2002.
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593